CLINICAL TRIAL: NCT01457521
Title: PAIN CONTROL IN FIRST TRIMESTER MEDICAL ABORTION: A Randomized Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Collaborators: Society of Family Planning (Other); Family Planning Associates Medical Group, LTD (Other); Planned Parenthood of Greater New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1000
Record Dates: First submitted 2011-10-20; First posted 2011-10-24 (Estimated); Results first posted 2016-01-13 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2015-10

CONDITIONS: Pain
Keywords: pain; medical abortion
MeSH Terms: conditions — Pain | interventions — Ibuprofen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Therapeutic (Active Comparator): Ibuprofen
  Interventions: Drug: Ibuprofen
- Prophylactic (Active Comparator): Ibuprofen
  Interventions: Drug: Ibuprofen

INTERVENTIONS:
Drug: Ibuprofen — Ibuprofen

SUMMARY:
This trial will compare two oral analgesic regimens in women undergoing first trimester medical abortion with mifepristone and misoprostol. The primary study outcome is pain.

DETAILED DESCRIPTION:
This trial will compare two oral analgesic regimens in women undergoing first trimester medical abortion with mifepristone and misoprostol. The primary study outcome is pain. Secondary objectives include comparing the regimens for the total amount of ibuprofen taken, use of other analgesics, vaginal bleeding, adverse events, successful completion of abortion, overall satisfaction with the abortion procedure.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with a gestational age of 63 days or less
* Desire a medical abortion with mifepristone and misoprostol

Exclusion Criteria:

- Have contraindications to ibuprofen

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Raymond, MD, MPH, Principal Investigator — Gynuity Health Projects
Locations (2):
- United States (2):
  - Family Planning Associates Medical Group, Chicago, Illinois
  - Planned Parenthood of New York City, Inc., New York, New York

REFERENCES:
- [Derived] Reynolds-Wright JJ, Woldetsadik MA, Morroni C, Cameron S. Pain management for medical abortion before 14 weeks' gestation. Cochrane Database Syst Rev. 2022 May 13;5(5):CD013525. doi: 10.1002/14651858.CD013525.pub2. PMID 35553047
- [Derived] Raymond EG, Weaver MA, Louie KS, Dean G, Porsch L, Lichtenberg ES, Ali R, Arnesen M. Prophylactic compared with therapeutic ibuprofen analgesia in first-trimester medical abortion: a randomized controlled trial. Obstet Gynecol. 2013 Sep;122(3):558-64. doi: 10.1097/AOG.0b013e31829d5a33. PMID 23921857

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylactic: Ibuprofen 800 mg starting 1 hour before the misoprostol dose and continuing every 4-6 hours for 48 hours regardless of pain, then as needed. The maximum dose is 3,200 mg per 24 hour period.
- Therapeutic: Ibuprofen 800 mg every 4-6 hours as needed starting at the onset of pain. The maximum dose is 3,200 mg per 24 hour period.
Period: Overall Study
Arm/Group | Prophylactic | Therapeutic
Started | 123 | 127
Completed | 111 | 117
Not Completed | 12 | 10

BASELINE CHARACTERISTICS:
Population: Inclusive of participants who provided follow-up data only
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylactic | Therapeutic | Total
Number analyzed (Participants) | 111 | 117 | 228
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 109 | 115 | 224
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 111 | 117 | 228
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: 11-point Visual Analog Scale for Pain
Description: Participant pain was assessed using an 11-point Visual Analog Scale for Pain. Scores ranged from 0 (no pain) to 10 (worst pain possible)
Time Frame: 1-2 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prophylactic | Therapeutic
Number analyzed (Participants) | 111 | 117
units on a scale | 7.1 (2.5) | 7.3 (2.2)

ADVERSE EVENTS:
Time Frame: 1-2 weeks (beginning the day of enrollment to the day the woman returned for follow-up after which her study participation concluded)
Arm/Group | Prophylactic | Therapeutic
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/127
Other Adverse Events (participants affected / at risk) | 0/123 | 0/127

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No